CLINICAL TRIAL: NCT06860698
Title: The Impact of Chronic E-Cigarette Usage on Microvascular Health
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20029023
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: E-Cig Use
Keywords: Microvascular Health
MeSH Terms: conditions — Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and breath condensate will be collected and stored and the department of Kinesiology and Health Sciences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic e-cigs users: Used e-cigarettes with nicotine (≥3 times/week for ≥6 months)
  Interventions: Other: E-cig use
- Never Users: Use of cigarettes or other tobacco products less than 50 times in their lifetime.
  Interventions: Other: E-cig use

INTERVENTIONS:
Other: E-cig use — Based on e-cigarette usage, participants will be divided into those who used e-cigarettes and those who did not use e-cigarettes

SUMMARY:
The study is focused on investigating the mechanisms involved in microvascular health in subjects that use e-cigarettes frequently. To explore microvascular health, different techniques and compounds. For one of the tests, iontophoresis, the drug's use will be stored and handled as described by the approved IND and non-IDS plan.

DETAILED DESCRIPTION:
Electronic cigarettes or e-cigarettes have become increasingly popular, due to their promotion as a healthy alternative to traditional tobacco cigarettes. However, there are large discrepancies of knowledge in understanding how these e-cigarettes affect the subjects health and the way their body uses oxygen. The overall goal of this study is to evaluate e-cigarettes usage on subjects health.

ELIGIBILITY:
e-Cig users arm

Inclusion Criteria:

* Between 18 and 29 years of age
* Used e-cigarettes with nicotine (≥3 times/week for ≥6 months)

Exclusion Criteria:

* 17 years old and younger or 30 years old or older.
* Former combustible tobacco user/ former smoker
* Use of cigarettes for 15 days or more in the past 60 days
* Use of other tobacco products (cigars, hookah, smokeless), marijuana and/or illicit or prescription drugs weekly or more frequently in the past 60 days
* Evidence of cardiovascular, pulmonary, renal, hepatic, metabolic, cerebral diseases or sleep disorders
* Disorder or use of medication that affects cardiopulmonary health
* Evidence of pregnancy or current nursing

Non e-Cig using arm

Inclusion

- Between 18 and 29 years of age

Exclusion

* 17 years old and younger or 30 years old and older
* Use of cigarettes or other tobacco products more than 50 times in their lifetime.
* Evidence of cardiovascular, pulmonary, renal, hepatic, metabolic, cerebral diseases or sleep disorders
* Disorder or use of medication that affects cardiopulmonary health
* Evidence of pregnancy or current nursing

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Chronic e-cigs users and never users that are between 18 and 29 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Endothelial dependent dilation | Participation is one week
  Endothelial-dependent dilation will be assessed using laser doppler speckle contrast in both groups through the intervention
Neurogenic response | Participation is one week
  Neurogenic response will be assessed using axon reflex in both groups through the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Paula Rodriguez Miguelez, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States